CLINICAL TRIAL: NCT00513994
Title: MQX-503 Applied to the Fingers vs. Nitroglycerin Ointment 2%, USP, Applied to the Chest: A Pharmacokinetic Comparison in Normal Subjects
Brief Title: MQX-503 vs Nitroglycerin Ointment: A Pharmacokinetic Comparison in Normal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediQuest Therapeutics (Industry)
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-002
Record Dates: First submitted 2007-08-07; First posted 2007-08-09 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Nitroglycerin; pharmacokinetics study of nitroglycerin containing treatments
MeSH Terms: interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator)
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Nitroglycerin — MQX-503 1%, a topical microemulsion of nitroglycerin 1% and Nitroglycerin Ointment 2%, USP
  Other Names: MQX-503, Nitro-Bid

SUMMARY:
The purpose of the study is to measure how much nitroglycerin or its metabolites may be found in the bloodstream when MQX-503 or an FDA approved Nitroglycerin ointment 2% USP is applied to the skin of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers 18 - 70 years of age.
* Subjects able to give written informed consent and comply with study requirements.
* Subjects willing and able to safely discontinue all current prescription therapies.
* Subjects who will agree not to participate in other clinical trials.
* Negative pregnancy test in fertile females and agreement to use effective contraception throughout the study.

Exclusion Criteria:

* Persons who would be put at risk by discontinuing prescription therapies.
* Subjects with a known allergy to nitroglycerin.
* Subjects who have a condition or issue that would adversely affect the application of study medication, study evaluations or the subject's ability to comply with the protocol.
* Subjects who recently experienced myocardial infarction, uncontrolled congestive heart failure, unstable angina, uncontrolled hypotension or uncontrolled hypertension.
* Subjects who have participated in a study of an investigational drug within two weeks of visit 1.
* Subjects who have screening lab values that are out of range or are considered clinically significant by the investigator.
* Subjects who have had major abdominal, thoracic, or vascular surgery within 6 months of visit 1.
* Subjects with non-epithelialized skin lesions or interfering skin conditions at the time of screening in the area where study medication is to be applied.
* Pregnant or nursing women.
* Women of childbearing potential who are unwilling to comply with the contraceptive requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2007-08; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary objective is the measurement and comparison of the levels of nitroglycerin and its metabolites in the blood of healthy human volunteers after a single topical dose of MQX-503 and a single topical dose of Nitroglycerin Ointment 2%, USP. | 8 hours

SECONDARY OUTCOMES:
A secondary objective is the observation of the volunteers for any adverse events | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adel Nada, M.D., Principal Investigator — Charles River Clinical Research
Locations (1):
- Charles River Clinical Services, Tacoma, Washington, United States